CLINICAL TRIAL: NCT01779479
Title: Randomized, Open-label, Phase II Study Comparing the Efficacy and the Safety of Cabazitaxel Versus Weekly Paclitaxel Given as Neo-adjuvant Treatment in Patients With Operable Triple Negative or Luminal B/HER2 Normal Breast Cancer (GENEVIEVE)
Brief Title: Efficacy and Safety of Cabazitaxel Versus Weekly Paclitaxel as Neo-adjuvant Treatment in Patients With Triple Negative or Luminal B/HER2 Normal BC (GENEVIEVE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 74; 2012-003330-16 (EudraCT Number)
Record Dates: First submitted 2013-01-25; First posted 2013-01-30 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2016-02

CONDITIONS: Primary Breast Cancer
Keywords: German Breast Group; GBG Forschungs GmbH; GBG; GBG 74; Genevieve; Breast Cancer; Primary Breast Cancer; Cabazitaxel; Paclitaxel; neo-adjuvant; triple negative; luminal B
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabacitaxel (Experimental)
  Interventions: Drug: Cabacitaxel
- Paclitaxel (Active Comparator)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Cabacitaxel — Cabazitaxel 25 mg/m² i.v. (Day 1) every 3 weeks (cycle) as 1-hour i.v infusion for a total of up to 4 cycles over a maximum total treatment period of 15 weeks before surgery
  Arms: Cabacitaxel
Drug: Paclitaxel — Paclitaxel 80 mg/m² as 1-hour i.v infusion. Patients will receive weekly (Days 1, 8, 15) paclitaxel administrations for a maximum of 12 infusions for a maximum of 4 cycles over a maximum total treatment period of 15 weeks before surgery (1 cycle = 3 weeks).
  Arms: Paclitaxel

SUMMARY:
Cabazitaxel is a new taxoid which promotes the tubulin assembly in vitro and stabilizes microtubules against cold-induced depolymerization as efficiently as docetaxel and was selected for development based on a better antiproliferative activity on resistant cell lines than docetaxel. It has shown superior survival against mitoxantrone (MTX) plus prednisone in docetaxel pre-treated hormone refractory metastatic prostate cancer patients leading to registration of the compound. It showed a favorable toxicity profile with an interestingly low rate of alopecia. In the Genevieve study it will be compared against weekly paclitaxel which is currently most widely used treatment of breast cancer patients. A head-to-head comparison in the neoadjuvant setting will allow a rapid and precise comparison of efficacy and tolerability of cabacitaxel versus paclitaxel to decide in how far further development of this taxoid in breast cancer is reasonable.

DETAILED DESCRIPTION:
Primary Objective To compare the pathologic complete response (pCR) rate in the breast (ypT0/is ypN0/+) in patients with operable Triple Negative or luminal B/HER2 normal breast cancer treated with either cabazitaxel or weekly paclitaxel.

Secondary Objective To assess

* pCR rates per arm separately for the stratified subpopulations.
* Objective response rate (ORR) in the breast according to WHO criteria.
* pCR rate defined as ypT0 ypN0.
* pCR rate defined as ypT0/is ypN0.
* pCR rate in the axillary lymph nodes (ypN0).
* To determine the pCR rate and local recurrence free survival (LRFS) in patients with a clinical complete response (cCR) and a negative core biopsy before surgery.
* Breast conservation surgery rate.
* To assess the toxicity (NCI CTCAE V4.03) and compliance in both arms.
* Invasive loco-regional recurrence free survival (LRRFS), distant-disease-free survival (DDFS), invasive disease-free survival (IDFS), and overall survival (OS).
* To explore the biomarkers and profiles potentially predicting response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study according to local regulatory requirements prior to beginning specific protocol procedures.
* Complete baseline documentation must be sent to GBG Forschungs GmbH.
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration alone is not sufficient. Incisional biopsy is not allowed. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* Tumor lesion in the breast with a palpable size of >= 2 cm or a sonographical size of >= 1 cm in maximum diameter. The lesion has to be measurable in two dimensions, preferably by sonography.
* Patients must be in the following stages of disease: cT3 or cT2 or cT1c and cN+ or cT1c and pNSLN+.
* In patients with multifocal or multicentric breast cancer, the largest lesion should be evaluated.
* Centrally confirmed triple negative or luminal B/HER2-normal subtype. ER- and PgR-negative defined as <1% stained cells. HER-2 negative defined as IHC 0+, 1+ or IHC 2+ and FISH/SISH/CISH (ratio <2.0) negative. Luminal B defined as ER and/or PgR + and > 14% Ki-67 stained cells. The formalin-fixed, paraffin-embedded (FFPE) breast tissue block from the diagnostic core biopsy has therefore to be sent to the Dept. of Pathology at the Charité, Berlin prior to randomization.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0 or 1 (see Appendix A).
* Laboratory requirements: Hemoglobin > 9.0 g/dL, Absolute neutrophil count > 1.5 x 109/L, Platelet count > 100 x 109/L, AST/SGOT and/or ALT/SGPT < 2.5 x ULN; Total bilirubin < 1.0 x ULN, Serum creatinine < 1.5 x ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance < 60 mL/min should be excluded (see Appendix 2 for formula).
* Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential.
* Complete staging work-up within 3 months prior to randomization. All patients must have bilateral mammography, breast ultrasound (<= 21 days), breast MRI (optional), chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRI, and bone scan done. In case of positive bone scan, bone X-ray is mandatory. Other tests may be performed as clinically indicated.
* Patients must be available and compliant for central diagnostics, treatment and follow-up.

Exclusion Criteria:

* Any prior treatment for primary breast cancer including radiation therapy
* History of ipsi/ or contra-lateral invasive breast cancer
* Locally advanced disease including N3 and metastatic disease
* Patients in the following stages of disease are not allowed: cT4
* Prior malignancy without being disease-free for more than 5 years (except carcinoma in situ of the cervix or other in situ cancer (e.g. bladder cancer) and adequately treated basal cell carcinoma of the skin.
* Clinically significant (i.e. active) cardiovascular disease, including cerebrovascular accident (≤6 months before enrolment), myocardial infarction, arterial thrombotic events (≤6 months before enrolment), unstable angina pectoris, New York Heart Association (NYHA) ≥ grade 2 congestive heart failure and/or hypertension, serious cardiac arrhythmia requiring medication during the study and that might interfere with regularity of the study treatment, or not controlled by medication
* Any severe acute or chronic medical condition which could impair the ability of the patient to participate to the study or to comply with the study procedures or interfere with interpretation of study results (such as significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures).
* Active infection.
* Sex hormones. Prior treatment must be stopped before study entry.
* Inability and unwillingness to comply with study visits, treatment, testing, and to comply with the protocol.
* Administration of any live virus vaccine within 8 weeks preceding study entry.
* Use of any investigational agent within 30 days of administration of the first dose of study drug or concurrent treatment on another clinical trial
* Requirement for radiation therapy concurrent with study anticancer treatment. Patients who require breast or chest wall radiation therapy after surgery are eligible
* Pregnancy or breastfeeding women
* Patients with childbearing potential who do not agree to use accepted and effective method of contraception (barrier methods, intrauterine contraceptive devices, sterilization) during the study treatment period and following a period of 6 months after the last study drug administration.
* History of hypersensitivity (grade ≥ 3) to polysorbate 80 or any study drugs or excipients
* Concurrent or planned treatment with potent strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a two-week wash-out period is necessary for patients who are already on these treatments) (see Appendix 3)
* Contraindications to the use of corticosteroid treatment
* Symptomatic peripheral neuropathy grade ≥ 2 (National Cancer Institute Common Terminology Criteria [NCI CTCAE] v.4.03).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | 15 months

SECONDARY OUTCOMES:
pathologic complete response (pCR) rate separately for subpopulations | 15 months
  pathologic complete response (pCR) rate separately for stratified subpopulations
Objective response rate (ORR) | 15 months
pCR rate defined as ypT0 ypN0 | 15 months
pCR rate defined as ypT0/is ypN0 | 15 months
pCR rate in the axillary lymph nodes (ypN0) | 15 months
pCR rate in patients with a clinical complete response (cCR) | 15 months
  To determine the pCR rate in patients with a clinical complete response (cCR) and a negative core biopsy before surgery
local recurrence free survival (LRFS) in patients with a clinical complete response (cCR) | 15 months
  To determine the local recurrence free survival (LRFS) in patients with a clinical complete response (cCR) and a negative core biopsy before surgery
Breast conservation surgery rate | 15 months
Toxicity | 15 months
  To assess the toxicity (NCI CTCAE V4.03) in both arms.
Compliance | 15 months
  To assess compliance in both arms.
Invasive loco-regional recurrence free survival (LRRFS) | 15 months
Distant-disease-free survival (DDFS) | 15 months
Invasive disease-free survival (IDFS) | 15 months
Overall survival (OS) | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, Prof. Dr., Principal Investigator — Luisenkrankenhaus Düsseldorf
Locations (1):
- Luisenkrankenhaus, Düsseldorf, Germany

REFERENCES:
- [Result] Kummel S, Paepke S, Huober J, Schem C, Untch M, Blohmer JU, Eiermann W, Gerber B, Hanusch C, Hilfrich J, Jackisch C, Schneeweiss A, Denkert C, Engels K, Klare P, Fasching PA, von Minckwitz G, Burchardi N, Loibl S. Randomised, open-label, phase II study comparing the efficacy and the safety of cabazitaxel versus weekly paclitaxel given as neoadjuvant treatment in patients with operable triple-negative or luminal B/HER2-negative breast cancer (GENEVIEVE). Eur J Cancer. 2017 Oct;84:1-8. doi: 10.1016/j.ejca.2017.06.037. Epub 2017 Jul 30. PMID 28768217